CLINICAL TRIAL: NCT05628155
Title: MAÏA - MAintain the Level of Independence Through Alimentation
Acronym: MAÏA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35RC21_9884_MAÏA
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Nursing Homes; Clinical Trial; Food
Keywords: elderly; nursing homes; omega-3 polyunsaturated fatty acids; malnutrition; sarcopenia.
MeSH Terms: conditions — Malnutrition; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral diet including n-3 PUFA intake (Experimental): Oral diet covering the nutritional requirements in macronutrients as recommended for people over 65 years of age (ANSES, 2019) and including intakes of n-3 PUFAs corresponding to the recommendations for people over 65 years of age
  Interventions: Other: Oral diet including n-3 PUFA intake
- Control (No Intervention)

INTERVENTIONS:
Other: Oral diet including n-3 PUFA intake — menus to cover the recommended intake of n-3 PUFAs (ALA =1% of total energy intake, i.e. 2.1 g/d, and EPA+DHA = 500 mg/d) (n-3 PUFA MENU), based on mass-market products that guarantee the n-3 PUFA RDAs and are available from the catering sector
  Arms: Oral diet including n-3 PUFA intake

SUMMARY:
Malnutrition has serious consequences: increased risk of falls, hospitalization and mortality. Malnutrition may accompany or aggravate another geriatric syndrome. The loss of muscle mass and function, called "sarcopenia" can itself lead to a loss of physical activity and therefore of independence.

It has been reported that changes in the quantity or quality of food intake could influence the onset or progression of sarcopenia. Thus, an optimized oral diet covering the energy and protein needs of the elderly people living in a nursing home is a key element of the malnutrition prevention strategy. It could help slow down the loss of independence and have a direct impact on the occurrence of the complications mentioned above, and therefore on the use of care.

In the elderly, as in the general population, the consumption of linoleic acid (LA), precursor of the omega 6 line, is too high, and that of alpha-linolenic acid (ALA), precursor of the omega 3 line, insufficient. The French National Institute against Cancer (INCA) 3 survey results indicate for the 65-79 year old population average ALA intakes of 0.9 g/d whereas the recommendation is 2 g/d. The same is true for long-chain n-3 PUFAs (eicosapentaenoic acid (EPA), docosahexaenoic acid (DHA)).

There are currently no recommendations specifically concerning nursing home populations. Only recommendations for non-frail people, over the age of 65, exist (ANSES, 2019). Experts recommend maintaining or even slightly increasing the consumption of portions of meat, eggs, fish, fruits and vegetables and dairy products.

In the elderly, as in adults, an imbalance of n-6/n-3 PUFA intake or insufficient n-3 PUFA intake could facilitate the occurrence of cardiovascular diseases and certain cancers. The possible prevention of other pathologies more specific to the elderly, such as degenerative diseases, makes the consumption of n-3 PUFAs relevant in this population.

Our approach aiming to cover the recommended dietary allowances (RDA) of n-3 PUFAs via the oral diet is therefore very original.

An oral diet containing these different sources of fatty acid intake, of various origins, and other essential nutrients for the elderly, would have the advantage of meeting the nutritional objectives on the one hand, and of offering a wide range of tastes, flavors, and texture, allowing to optimize their consumption by nursing home residents, on the other hand. No study has yet evaluated the benefits of n-3 PUFA intake in dependent elderly people residing in nursing homes, moreover, using loss of independence as the main endpoint.

The main objective of the trial is to evaluate the effect of an everyday diet containing n-3 PUFA intakes corresponding to the RDA (population > 65 years) compared to the usual diet (therefore uncontrolled) on the evolution of the loss of independence at 2 years of nursing home residents.

DETAILED DESCRIPTION:
Prospective, controlled, randomized, multicentre, open-label clinical study comparing two groups of residents:

* "Control" group: nursing home residents will receive an oral diet covering their nutritional needs in macronutrients as recommended for people over 70-65 years of age.
* "Intervention" group: nursing home residents will receive an oral diet covering their nutritional needs in macronutrients as recommended for people over 65-70 years of age and including n-3 PUFA intake corresponding to the RDAs for people over 65 years.

Residents will be included in clusters corresponding to the nursing homes in which they reside.

The intervention will be delivered "at the nursing home level", i.e. all the residents included in the same nursing home will belong to the same "control" or "intervention" group.

Notes: Note that a randomization of residents across the individual residents was not possible from a logistical point of view in a context of collective feeding in an institution.

Actimetry analyzes as a marker of frailty. The investigators will conduct an ancillary study of actimetry analysis, on a sub-population of 60 residents (n=30 per group), in order to quantify physical activity and try to identify a possible trajectory of frailty that The investigators can correlate to the studied endpoints. To do this, the investigators will have a device consisting of an accelerometer and a barometer which will be positioned in a case around the neck (pendant) or failing that - if the resident expresses a preference - on the wrist (bracelet) to monitor participants' activities for 24 months. The nursing homes concerned will be selected for their proximity to Rennes and the homogeneity of the physical activities routinely offered to residents. The measures will be performed one week per month for 24 months.

Main judgment criterion: Measurement of the level of independence by the ADL-LFS (Activities of Daily Living - Long Form Score) at 2 years from the RAI-MDS 3.0 questionnaire (Resident Assessment Instrument Minimum Dataset) LTCF (Long-Term Care Facilities).

Secondary endpoints:

Evaluate the effect of an everyday diet containing n-3 PUFA intakes corresponding to the RDA (population > 65 years) compared to the usual diet (therefore uncontrolled) on the following endpoints:

1. The evolution of anthropometric criteria and malnutrition
2. The risk of falling
3. The risk of an infection occurring
4. The evolution of the quality of life
5. Mortality
6. Healthcare consumption (hospitalizations and visits to the emergency room)
7. In a sub-population of 60 residents (n=30 per group) randomly selected among the participants of a few volunteer nursing homes and meeting the inclusion and non-inclusion criteria of the study.

   * The evolution of the quality of physical and sporting activity
   * The evolution of the quality of sleep

   Organic:
8. The biological profile of blood fatty acids and concentrations of ALA, EPA, DPA, DHA in red blood cells
9. Micro-CRP and albumin
10. Evaluation of the cost of implementing the nutritional intervention from the perspective of nursing homes vs the clinical benefits

ELIGIBILITY:
Inclusion Criteria:

* Residents in permanent accommodation in participating nursing homes during the inclusion period;
* Residents in accommodation in nursing homes with similar catering services and who are not supplied with Bleu Blanc Coeur® food or who are supplied with at most 2 BBC products per week;
* Affiliation to a social security scheme;
* Consent signed by the resident or the person in charge of the representative

Exclusion Criteria:

* ADL-LFS score on inclusion >19;
* Exclusive enteral nutrition;
* Protection of effective justice;
* Lack of understanding of the French language;
* Estimated life expectancy of less than 12 months on inclusion, estimated by the attending physician or, if there is one, the nursing home physician.
* Only for the ancillary actimetry study: residents under guardianship or unable to self-manage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
independence level | at 2 years
  Measurement of independence level of by the ADL-LFS (Activities of Daily Living - Long Form Score) at 2 years. The evaluation criterion used is the functional numerical scale from 0 to 28 (0 = independent, 28= total dependence)

CONTACTS AND LOCATIONS:
Overall Officials: Ronan THIBAULT, MD, PhD, Principal Investigator — Rennes University Hospital
Locations (1):
- Les jardins d'Hermine, Rennes, France